CLINICAL TRIAL: NCT02526095
Title: National Oesophageal and Gastric Carcinomas Data Base Construction: the FREGAT (French EsoGastric Tumours) Data Base
Brief Title: The French EsoGastricTumours Data Base
Acronym: FREGAT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: French Eso-Gastric Tumors Working Group (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2013_33; 2013-A01281-44 (Other: ID RCB number, ANSM)
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Esophageal Disease
Keywords: Esophagus; Surgery
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study aims at evaluating the outcomes of gastrointestinal stromal tumor after surgery.

ELIGIBILITY:
Inclusion Criteria: Patient with

* esophageal cancer, gastric or gastroesophageal junction diagnosed biopsy , regardless of the subtype of cancer, tumor stage or treatment envisaged.
* Naive treatment for this cancer,
* Naive treatment for this cancer , failing that received neoadjuvant treatment ,
* Male or female ≥ 18 years.
* social protection scheme .
* sign a free and informed consent for blood sampling , the different questionnaires and the collection of patient information.

Exclusion Criteria:

Male or female aged ( e) under 18 years.

* Private person of liberty or under supervision (including guardianship ) .
* People who do not speak French.
* Major Nobody unable to consent .
* Patient FREGAT already included in the base.
* Patient Refusal .

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with gastroesophageal cancer diagnosed and treatment-naïve, if not receiving neoadjuvant treatment in a participating center will be included after acceptance and signature of consent, whether operated or not, whatever histologic type, tumor stage, and the therapeutic strategy.
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2014-06; Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
DIsease free survival | 5 year disease free survival

SECONDARY OUTCOMES:
overall survival | 5 year overall survival
recurrence rate | 5 year recurrence rate
Total number of patients with complications | from the time between inclusion and occurrence of the event, for the duration of 3 years
Total number of complications | from the time between inclusion and occurrence of the event, for the duration of 3 years
Death | from the time between inclusion and occurrence of the event, for the duration of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Piessen, MD, PhD, Study Director — University Hospital, Lille
Locations (31):
- France (31):
  - Chu Amiens Picardie, Amiens
  - Chru Besancon, Besançon
  - Hu Paris Site Avicenne Aphp, Bobigny
  - Chu de Caen Normandie, Caen
  - Crlcc Francois Baclesse, Caen
  - Hopital Estaing - Chu63 - Clermont Ferrand, Clermont-Ferrand
  - Hu Paris Nord Site Louis Mourier Aphp, Colombes
  - Hopital Le Bocage Chru Dijon, Dijon
  - Chu de Grenoble Alpes, Grenoble
  - Hop Claude Huriez Chu Lille, Lille
  - Clcc Oscar Lambret Lille, Lille
  - C H U Dupuytren Limoges, Limoges
  - Hospices Civils de Lyon (Pierre Bénite,Edouard Herriot, La Croix Rousse), Lyon
  - Aphm Hopital Nord, Marseille
  - Hopital St Eloi Chu Montpellier, Montpellier
  - Icm - Montpellier, Montpellier
  - Chu de Nantes :Site Hôtel-Dieu- Hme, Nantes
  - Chu Nimes, Nîmes
  - Hu Est Parisien Site St Antoine Aphp, Paris
  - Hu Paris Centre Site Cochin Aphp, Paris
  - Hu Paris Sud Site Kremlin Bicetre Aphp, Paris
  - Hu Saint Louis Site Saint Louis Aphp, Paris
  - Hopital Haut-Leveque - Chu - Pessac, Pessac
  - Hopital Robert Debre Chu Reims, Reims
  - Chru Rennes Site Pontchaillou, Rennes
  - Hopital Charles Nicolle Chu Rouen, Rouen
  - Hus/Hop Hautepierre, Strasbourg
  - Hopital Purpan Chu, Toulouse
  - Chu de Tours, Tours
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mariette C, Renaud F, Piessen G, Gele P, Copin MC, Leteurtre E, Delaeter C, Dib M, Clisant S, Harter V, Bonnetain F, Duhamel A, Christophe V, Adenis A; Fregat Working Group. The FREGAT biobank: a clinico-biological database dedicated to esophageal and gastric cancers. BMC Cancer. 2018 Feb 6;18(1):139. doi: 10.1186/s12885-018-3991-8. PMID 29409462
- See also: Related Info — https://www.fregat-database.org/